CLINICAL TRIAL: NCT02396277
Title: Structural and Functional Nerve Changes Following Immobilisation After Distal Radius Fracture - a Pilot Study (NRP)
Acronym: NRP
Status: Withdrawn | Type: Observational
Why Stopped: Due to limited resources
Sponsor: University of Tromso (Other)
Responsible Party: Sponsor
Other Study IDs: 2014/86 (REK)
Record Dates: First submitted 2015-03-17; First posted 2015-03-24 (Estimated); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Colles' Fracture; Distal Radius Fracture
MeSH Terms: conditions — Colles' Fracture; Wrist Fractures | interventions — Immobilization

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Immobilization — This is not an intervention study; but the patients are subjected to immobilization with a cast as part of a regular clinical treatment for distal radius fracture.

SUMMARY:
Immobilization after radius fracture seems to increase the risk of developing a Complex regional pain syndrome (CRPS), a condition associated with pain, increased skin sensitivity and reduced epidermal nerve density.

The purpose of the study is to determine whether 5-week immobilisation leads to functional and structural sensory changes, and whether the changes are associated with persistent pain. The investigators plan an explorative, pilot study on six consenting patients immobilised after a distal radius fracture.

The baseline measurements will be recorded at the day of or the day after trauma: Demographics, psychological and physical comorbidity, pain characteristics and intensity, hand function, health related quality of life (HRQOL), quantitative sensory testing will be recorded while skin biopsies are analyzed for epidermal nerve fiber density. Following variables such as pain characteristics and intensity, hand function, health related quality of life, quantitative sensory testing and skin biopsies will be reassessed when the cast is removed and two months later.

DETAILED DESCRIPTION:
Distal radius fracture is a prevalent injury, affecting 15.000 cases in Norway every year. About 5% of these patients suffer from longlasting pain and some develop a serious and chronic CRPS. Patients subjected to hand surgery frequently report pain one month after cast removal, and further examinations have revealed vascular and trophic changes, and increased sensitivity to pressure and cold as well as elevated skin levels of proinflammatory mediators.

Long term immobilization seems to increase the risk of developing CRPS symptoms. In a Danish study healthy volunteers demonstrated increased hyperalgesia to cold and mechanical stimuli even after 4-week immobilization which may indicate an early change in the nerve function.

In CRPS patients skin biopsies have demonstrated reduced epidermal nerve fiber density, but such data are lacking after radius fracture and during early stage of CRPS.

The purpose of this explorative, observational, pilot study is to investigate whether radius fracture followed by 5-week of immobilization, leads to functional and structural changes of the sensory system which are reversed after remobilization and whether the sensory changes are associated with persistent pain.

Our hypotheses are: 1) Patients with an immobilised arm following a radius fracture develops a) early cutaneous hypersensitivity (hyperalgesia and allodynia) for mechanical og thermal stimuli and b) reduced epidermal nerve fiber density.

2) The changes of the sensory system are reversed after 2-month remobilization. 3) The functional and structural changes are correlated with patient reported outcome measures (PROM) such as disability of arm, shoulder and hand (DASH), with pain intensity (NRS), duration of the pain and HRQOL .

Eligible patients will be included throughout 2015, and results will be analyzed within December 2015.

Measurements:

Self reported: Demographics (age, gender, civil state, education, working status, social security benefits) and clinical data of comorbidity, pain characteristics (DN4) and intensity (NRS), blood pressure, smoking /other kind of nicotine use, pain medication, and assessment scales for mental distress (HSCL 25), pain catastrophizing (PCS), hand function (DASH), and HRQOL (EQ5D).

Examinations: Quantitative sensory testing (tactile and thermal stimuli) and skin biopsies are carried out 10 cm proximal to fracture line on the dorsum of the affected arm. Measurements for predictor analyses will only be performed at baseline while outcome measurements will be performed prior to and just after removal of the cast as well as two months later.

Statistical analyses:

Regression analyses will be performed to identify other predictors for the changes in sensory nervous system including blood pressure, smoking /other kind of nicotine use, medication, age, gender, and comorbidity. Longitudinal analyses of numerical outcome (ANOVA repeated measurement) will be carried out for outcome measurements such as pain intensity,hand function, HRQOL, sensory thresholds and epidermal nerve fiber density.

ELIGIBILITY:
Inclusion Criteria:

* Consent competence
* Acute stable distal radius fracture (less than 48 hours)
* Allocated to conservative treatment with 5-week immobilization

Exclusion Criteria:

* Comorbidity which may prevent completion of the study
* Serious and progressive disease
* Chronic shoulder disease with limited ROM and function.
* Sign peripheral nerve injury in the upper extremities
* Polyneuropathy
* Demyelination disease
* Diabetes mellitus
* Anticoagulants including acetyl salicylic acid (ASA)
* Allergy to local anesthetics

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to the Emergency Clinic at The University Hospital in North Norway Tromso day time
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in nerve fiber density at five weeks | From baseline to five weeks after injury
  ANOVA repeated measurements based on repeated skin biopsies
Changes from baseline in sensitivity to thermal and tactile stimuli at five weeks | From baseline to five weeks after injury
  ANOVA repeated measurements based on repeated sensory quantitative testing

SECONDARY OUTCOMES:
Changes from five weeks in nerve fiber density at 13 weeks | From five weeks to 13 weeks after injury
  ANOVA repeated measurements based on results from repeated skin biopsies
Changes from five weeks in sensitivity to thermal and tactile stimuli at 13 weeks | From five to 13 weeks after injury
  ANOVA repeated measurements based on sensory quantitative testing
Correlation between changes in pain intensity and changes in nerve fiber density | From baseline to 13 weeks
  Statistical regression analyses based on repeated assessments of self reported pain intensity and skin biopsies
Correlation between changes in pain intensity and changes in sensitivity to thermal and tactile stimuli | From baseline to 13 weeks
  Statistical regression analyses based on repeated assessments of self reported pain intensity and quantitative sensory testing
Changes from baseline (preinjury) in disability of arm, shoulder and hand are correlated with changes in pain intensity at five and 13 weeks | From baseline to 13 weeks
  Statistical regression analyses based on repeated self reports of pain intensity and DASH
Changes from baseline (preinjury) HRQOL are correlated with changes in pain intensity at five and 13 weeks | From baseline to 13 weeks
  Statistical regression analyses based on repeated self reports of pain intensity and HRQOL (EQ5D)

CONTACTS AND LOCATIONS:
Overall Officials: Gunnvald Kvarstein, PhD, Study Chair — University of Tromso
Locations (1):
- University Hospital of North Norway, Tromsø, Norway